CLINICAL TRIAL: NCT07403851
Title: Effect of Scanning Technology on the Accuracy of Digitally Customized Intraradicular Attachments: A Cross Overstudy
Brief Title: Effect of Scanning Technology on the Accuracy of Digitally Customized Intraradicular Attachments
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Afnan Gamal Mohamed Qamar, Teaching assistant in removable prosthodontic department, October 6 University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Effect of Scanning Technology
Record Dates: First submitted 2025-09-29; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-09

CONDITIONS: Scanning Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Active Comparator): Indirect scanning by desktop scanner (for the conventional impression)
  Interventions: Device: 3 shape desktop scanner
- Group II (Experimental): Intraoral scanning by Intraoral scanner A
  Interventions: Device: SHINING 3D intraoral scanner
- Group III (Experimental): Intraoral scanning by Intraoral scanner B
  Interventions: Device: Planmeca Emerald S intraoral scanner

INTERVENTIONS:
Device: 3 shape desktop scanner — Scanning of intra-radicular impression by desktop scanner
  Arms: Group I
Device: SHINING 3D intraoral scanner — Direct scanning of the intra-radicular canal by Intraoral scanner A
  Arms: Group II
Device: Planmeca Emerald S intraoral scanner — Direct scanning of the intra-radicular canal by Intraoral scanner B
  Arms: Group III

SUMMARY:
This study aims to evaluate the accuracy of intra-radicular attachments fabricated by direct scanning using three different scanners in vivo. The primary outcome will be the accuracy of the fabricated attachments, while secondary outcomes will includepatient-reported comfort during procedure of taking intraradicular attachment conventional impression and direct scanning.

DETAILED DESCRIPTION:
The fabrication of intra-radicular attachments is a critical step in restoring endodontically treated teeth. The accuracy of these restorations directly impacts their clinical performance, including retention, marginal fit, and long-term success. With advancements in digital dentistry, intraoral scanners (IOS) have become increasingly popular for direct scanning of intra-radicular preparations. However, the accuracy of these scanners varies depending on their technology, software, and clinical conditions

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-65 years.
2. Endodontically treated teeth requiring intra-radicular attachments.
3. Adequate oral hygiene .
4. Partially edentulous case ( Compromised remaining teeth that cannot serve as abutments for traditional RPD.
5. Periodontally Compromised Teeth: When some teeth have reduced bone support but can still be maintained as overdenture abutments with proper treatment.

Exclusion Criteria:

1. Severely Compromised Remaining Teeth: If the remaining teeth have poor prognosis due to extensive decay or severe periodontal disease.
2. Severe Bone Loss Around Abutment Teeth: If the remaining teeth do not provide adequate support, they may fail early, leading to additional complications.
3. Severe Malocclusion: Where occlusal discrepancies make overdenture placement difficult.
4. Limited inter-arch Space: cann't accommodate the overdenture components. 5 .Poor Oral Hygiene: increase the risk of decay or periodontal issues in retained abutments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy | Immediately after scanning.
  measure accuracy between the dimension of the prepared canal gained by intra-radicular impression and the dimension of the prepared canal directly by two different types of intraoral scanners

SECONDARY OUTCOMES:
Patient-reported comfort | Immediately after impression taking and scanning.
  Patient-reported comfort (assessed via a Likert scale questionnaire) Scaled from 0-100 The highest score means excellent The lowest score means unsatisfactory